CLINICAL TRIAL: NCT02682641
Title: Multicentric Phase II Trial to Evaluate the Efficacy and Safety of Ibrutinib in Combination With Rituximab in Patients With Indolent Clinical Forms of Mantle Cell Lymphoma
Brief Title: Ibrutinib in Combination With Rituximab in Patients With Indolent Clinical Forms of MCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELTAMO-IMCL-2015; 2015-004158-17 (EudraCT Number)
Record Dates: First submitted 2016-01-18; First posted 2016-02-15 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IBRUTINIB + RITUXIMAB (Experimental): Subjects will receive the ibrutinib in combination with rituximab according to the following schedule:
  * Ibrutinib 560 mg daily po until disease progression or unacceptable toxicity. In case of sustained negative MRD (at least for 6 months) after 2 years of continuous therapy, ibrutinib will be discontinued.
  * Rituximab 375 mg/m2 iv day 1,8, 15 and 22 (cycle 1). Rituximab 375 mg/m2 iv, day one of every cycle 3, 5, 7 and 9.
  Interventions: Drug: IBRUTINIB; Drug: Rituximab

INTERVENTIONS:
Drug: IBRUTINIB — Ibrutinib 560 mg daily po for 28 days (cycle one). Continuous cycles until disease progression or unacceptable toxicity.
  Other Names: Imbruvica
Drug: Rituximab — Rituximab 375 mg/m2 iv day 1,8, 15 and 22 (cycle 1, 4 doses). Rituximab 375 mg/m2 iv, day one of every other cycle for 4 doses (cycle 3, 5, 7 and 9).

SUMMARY:
Phase II study with a two-stage design to evaluate efficacy and safety of ibrutinib in combination with rituximab (I+R) in untreated patients with indolent clinical forms of MCL.

An extensive biological study will be conducted in order to further characterize this population of MCL patients and evaluate the response obtained with the mutational profile of the tumor.

DETAILED DESCRIPTION:
Patients with mantle cell lymphoma (MCL) have a median survival of 3-5 years despite treatment. Indeed, the best therapeutic approach for different patients with MCL remains to be established, coexisting different options of immunochemotherapy regimes which may include autologous transplantation in first-line treatment or rituximab maintenance.

Moreover, last years MCL starts to be recognized as a heterogeneous disease both from biological and clinical stand points. For instance, MCL cases with a non-nodal clinical presentation, usually have distinctive biological features such as SOX-11 negativity, hypermutated IGHV genes and a low number of genetic lesions associated. The outcome of these cases is much more favourable compared to conventional MCL, reaching median survivals over 7 to 10 years even receiving less intensive treatments. In addition to that, up to 30% of the patients with newly diagnosed MCL can be safely deferred from initial therapy until progression . Therapeutic abstention may be prolonged for more than one year in 50% of cases. These patients usually show longer survivals from the start of treatment compared to patients immediately treated after diagnosis. Therefore, all these observations indicate that there are indolent clinical forms in MCL, so its clinico-biological identification is crucial to tailor treatment appropriately. However, at present there is no consensus on the diagnostic criteria or treatment recommendations in cases of indolent MCL. This results in difficulties for the identification of these forms in the clinical practice as well as with a certain therapeutic in definition, as indolent forms of MCL can be treated either with therapeutic abstention until progression or receive immediate treatment with conventional or more intensive immuno-chemotherapy regimes, which may even include an autologous hematopoietic stem cell transplantation. With the emergence of new biological agents in the therapeutic arsenal of MCL arises the question whether a completely different approach with new drugs and chemotherapy-free could be more appropriate in selected subsets of patients such as indolent MCL forms.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with confirmed diagnosis of Mantle Cell Lymphoma (World Health Organization Classification, WHO 2008). Classical, small-cell variants and marginal-zone variants can be included.
2. Age 18 years or older.
3. Subjects must not have received any prior therapies (excluding diagnostic splenectomy).
4. Asymptomatic patients.
5. Ann Arbor clinical stages I-IV.
6. Eastern Cooperative Oncology Group (ECOG) performance status <2 (0-1).
7. Subjects with a non-nodal MCL presentation with mainly bone marrow or peripheral blood involvement.
8. Other asymptomatic clinical presentations are acceptable in case of low tumor burden, including nodal MCL with lymph node enlargement ≤3 cm in the maximum diameter and with low proliferation index (Ki-67 ≤ 30%).
9. The following laboratory values at screening: a) Neutrophil count ≥ 1×10e9/L, Hemoglobin level ≥ 100 g/L or platelet count ≥100×10e9/L; b) Transaminases (AST and ALT) ≤ 3 x ULN. c)Total bilirubin ≤1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin; d) Creatinine ≤ 2 x ULN or calculated creatinine clearance ≥ 40 mL/min/1.73 m2.
10. Stable disease without evidence of clinical progression criteria for at least 3 months. Patients in prolonged therapeutic abstention may be included.
11. Women of childbearing potential and men who are sexually active must be practising a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
12. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
13. Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

1. Aggressive histological variants: blastic and pleomorphic variants (blastoid).
2. Proliferation index measured by Ki-67 > 30%.
3. B-cell monoclonal lymphocytosis with MCL phenotype
4. Eastern Cooperative Oncology Group (ECOG) performance status ≥2. Presence of B symptoms or any relevant symptoms related to the MCL.

6. Nodal clinical forms with lymph node enlargement >3 cm (maximum diameter). 7. Cytopenias attributable to MCL: Neutrophil count < 1×10e9/L, Hemoglobin level < 100 g/L or platelet count < 100×10e9/L.

8. Organ dysfunction related to MCL including creatinine level > 2 x ULN or altered liver biochemistry (> 3x ULN).

9. Gradual increase in different determinations of serum LDH attributable to MCL that exceeds 20% of the ULN.

10. Known CNS infiltration. 11. Subjects with expected therapy requirement for MCL in a short time (< 3 months) 12. Patients with active hepatitis B or C infection or HIV infection. Positive test results for chronic HBV infection (defined as positive HBsAg serology) or positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing) will be excluded with the following exceptions. Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing or antiviral prophylaxis. Patients who have protective titers of hepatitis B surface antibody (HBsAb) after vaccination or prior but cured hepatitis B are eligible. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.

13. Anticoagulation requirement with vitamin K antagonists. 14. Past medical history of stroke or intracranial haemorrhage within 6 months prior to inclusion.

15. Required medication with strong CYP3A4/5 inhibitors 16. Any serious comorbidity that makes the patient unacceptable for receiving the treatment.

17. Concomitant or previous malignancies the last 2 years other than basal skin cancer or in situ uterine cervix cancer.

18. Pregnancy or lactation. 19. Major surgery within 4 weeks of inclusion. 20. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.

21. Vaccinated with live, attenuated vaccines within 4 weeks of randomization. 22. Uncontrolled systemic infection requiring intravenous (IV) antibiotics. 23. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05-18 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission | 12 months
  Percentage of patients who are alive and in complete response at 12 months from the date of treatment initiation. All patients will be evaluated with PET- CT and bone marrow biopsy at that time.

SECONDARY OUTCOMES:
Overall Response Rate (OR) | 12 months
  Including complete response and partial response according to the International Response Criteria for Non- Hodgkin Lymphoma
Progression Free Survival | 7 years
  Percentage of patients without progression of disease
Response Duration | 7 years
  Length of time between
Minimal residual disease (MRD) | within 12 months after initiation of study treatment
  Proportion of subjects who are MRD negative (ie, less than the lower limit of detection for the MRD assay).
Overall survival | 7 years
  Percentage of patients alive from first dose of treatment to end of follow-up.
Adverse Events (AEs), Serious Adverse Events (SAES) and Suspected Unexpected Serious Adverse Reactions (SUSARs) | 7 years
  Number of events classified according to the Common Toxicity Criteria of the National Cancer Institute (CTC AE V 4.03).
Score of the EORTC quality of life questionnaire QLQ-30 | 12 months
  Health related quality of life questionnaire
Secore of the FACT-LYM | 12 months
  Health related quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eva Giné, MD, Study Chair — Hospital Clinic of Barcelona
Locations (15):
- Spain (15):
  - Hospital Universitario Mútua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Clinico de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gine E, de la Cruz F, Jimenez Ubieto A, Lopez Jimenez J, Martin Garcia-Sancho A, Terol MJ, Gonzalez Barca E, Casanova M, de la Fuente A, Marin-Niebla A, Muntanola A, Gonzalez-Lopez TJ, Aymerich M, Setoain X, Cortes-Romera M, Rotger A, Rodriguez S, Medina Herrera A, Garcia Sanz R, Nadeu F, Bea S, Campo E, Lopez-Guillermo A. Ibrutinib in Combination With Rituximab for Indolent Clinical Forms of Mantle Cell Lymphoma (IMCL-2015): A Multicenter, Open-Label, Single-Arm, Phase II Trial. J Clin Oncol. 2022 Apr 10;40(11):1196-1205. doi: 10.1200/JCO.21.02321. Epub 2022 Jan 14. PMID 35030036